CLINICAL TRIAL: NCT00249444
Title: A Placebo Controlled Trial of Mirtazapine for Patients With Depression and Cocaine Dependence
Brief Title: Mirtazapine for Treating Cocaine Dependent Individuals Who Also Suffer From Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5086/6177R NIDA-09236-13; P50DA009236 (NIH); P50DA009236-13 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Cocaine Dependence; Depression
Keywords: cocaine dependence; mirtazipine
MeSH Terms: conditions — Cocaine-Related Disorders; Depression | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirtazapine (Active Comparator): Mirtazapine will be administered on a fixed-flexible schedule, with dose titrated up to 60 mg per day or the maximum tolerated dose.
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine
  Other Names: Remeron
  Arms: Mirtazapine
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
Many substance dependent individuals also suffer from depression. Past research suggests that antidepressant medication is helpful in treating such individuals. This study will determine the effectiveness of mirtazapine, an antidepressant medication, in treating cocaine dependent individuals who also suffer from depression. This study includes free treatment for cocaine dependence that includes medication and a behavioral intervention.

DETAILED DESCRIPTION:
Cocaine abuse and depression often occur together. Individuals suffering from both are usually not able to quit abusing cocaine. Past research conducted on alcohol dependent individuals also suffering from depression showed that these individuals were able to successfully quit drinking with the addition of an antidepressant medication. Mirtazapine is a medication currently used to treat depression. This study will evaluate the efficacy of mirtazapine, used in combination with behavioral therapy, in treating cocaine dependent individuals who also suffer from depression.

Participants in this 8-week trial will be randomly assigned to receive either mirtazapine or placebo. Prior to starting medication treatment, participants will undergo an initial 2-week phase consisting of psychosocial and behavioral therapy. The purpose of this lead-in phase is to achieve initial reduction or abstinence in cocaine use, while observing cocaine withdrawal symptoms and mood changes associated with depression. During these first 2 weeks, participants will attend three study visits each week, at which time they will participate in motivational interviews and cognitive behavioral relapse prevention therapy. During this phase, participants who successfully remain abstinent from cocaine use will be rewarded with high-value monetary vouchers.

Upon completing the lead-in phase, participants will be randomly assigned to receive either mirtazapine or placebo. Participants will attend study visits twice each week for 8 weeks. Mood and drug use will be evaluated at each study visit. Cognitive behavioral relapse prevention therapy will continue throughout the study. In addition, participants will earn low-value monetary vouchers contingent on cocaine abstinence.

At the end of Week 8, participants will enter the lead-out phase. At this time, those participants whose mood has significantly improved will be able to continue treatment for an additional 8 weeks. Participants whose mood has not shown improvement will be tapered off their assigned medication treatment and will be offered treatment with an alternative medication. Following completion of the lead-out phase, all participants will be referred for continuing care in the community.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current cocaine dependence
* Currently seeking treatment for cocaine dependence
* Used cocaine for at least one day per 2-week period in the month prior to study entry
* Meets DSM-IV criteria for current major depression or dysthymia syndrome
* Scores greater than 12 on the Baseline 21 Hamilton Depression Scale
* Ages 18-60

Exclusion Criteria:

* Meets DSM-IV criteria for past mania (e.g., bipolar disorder), schizophrenia, or any psychotic disorder other than transient psychosis due to drug abuse
* Scores less than 11 on the Baseline 21 Hamilton Depression Scale
* History of seizures
* History of an allergic reaction to mirtazapine
* Chronic organic mental disorder
* Current suicidal risks or any history of suicidal behavior
* Pregnant, breastfeeding, or unwilling to use an adequate method of contraception for the duration of the study
* Unstable physical disorders, including high blood pressure, acute hepatitis, or diabetes
* Coronary vascular disease as indicated by history, or suspected by abnormal electrocardiogram, or history of cardiac symptoms
* Cardiac conduction system disease, as indicated by an electrocardiogram QRS duration greater than 0.11
* History of failure to respond to a previous trial of mirtazapine
* Currently taking psychotropic medication
* Meets DSM-IV criteria for opioid or sedative-hypnotic dependence
* Meets DSM-IV criteria for alcohol dependence with evidence of clinically significant physiological dependence in need of medically supervised detoxification
* Current alcohol or marijuana dependence identified as the main problem for seeking treatment; individuals with alcohol or marijuana dependence (without significant physiological dependence) and cocaine dependence are eligible, as long as cocaine is identified as the primary substance problem for which they are seeking treatment
* History of neutropenia (< 500 granulocytes /cc) or Agranulocytosis (<500 granulocytes/cc) with fever, infection. Concurrent intake of medications with possible neutropenic effects: chlorpromazine, carbamazepine, clozapine, chemotherapeutic drugs, immunosuppressant medications, interferons, ganciclovir, protease inhibitors.
* Patients not able to meet attendance requirement of 4/6 visits during the lead-in period.
* Supplemental exclusion criteria for cold pressor test (CPT): history of frostbite, open cut or sore on foot to be immersed, history of Raynaud's phenomenon.
* Supplemental exclusion criteria for CPT: hypertension (BP less than or equal 140/90)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2006-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfrid Raby, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Research Foundation for Mental Hygiene, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: service website — http://www.stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a 2 week (no medication) lead-in period prior to randomization. To be randomized, patients had to attend at least 4 of 6 clinic visits, and submit at least 4 of 6 urine samples for toxicology during these two weeks. 86 participants were randomized.
Period: Overall Study
Arm/Group | Mirtazapine | Placebo
Started | 42 | 44
Completed | 30 | 29
Not Completed | 12 | 15
Not completed — Lost to Follow-up | 2 | 2
Not completed — non-compliant | 9 | 11
Not completed — Adverse Event | 1 | 1
Not completed — life event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirtazapine | Placebo | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (7.6) | 42.9 (8.4) | 42.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 37 | 34 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 17 | 29
  White | 16 | 11 | 27
  More than one race | 12 | 14 | 26
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Abstinence During Last Three Weeks of Study
Description: measured daily by self report and confimed by urine toxicology for 8 weeks of the trial or length of study participation
Time Frame: measured daily by self report and confimed by urine toxicology for 8 weeks of the trial or length of study participation
Measure: Number; unit: participants
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 42 | 44
participants | 5 | 9

2. Primary Outcome: Depression Score on Hamilton - Depression 25 Item
Description: Participants those who had a 50% decrease in HAM-D scores from baseline at end of study. The outcome measured is 50% drop in Hamilton score at week 8 or last week of study participation compared to baseline. We looked at the difference between baseline score and score at week 8 or last week of study participation.
Time Frame: End of 8 week study or last week of participation
Measure: Number; unit: participants
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 42 | 44
participants | 38 | 42

ADVERSE EVENTS:
Time Frame: during 2 week lead-in and 8 weeks of trial or course of study participation
Arm/Group | Mirtazapine | Placebo
Serious Adverse Events (participants affected / at risk) | 2/42 | 0/44
Other Adverse Events (participants affected / at risk) | 20/42 | 4/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirtazapine (N=42) | Placebo (N=44)
depression (Psychiatric disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirtazapine (N=42) | Placebo (N=44)
somnolence (General disorders) | 5 (5) | 0 (0)
weight gain (General disorders) | 9 (9) | 0 (0)
dizziness (General disorders) | 2 (2) | 1 (1)
restlessness (General disorders) | 1 (1) | 2 (2)
appetite increase (General disorders) | 5 (5) | 0 (0)
sweating (General disorders) | 1 (1) | 1 (1)
hypertension (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early cocaine responders were the most likely to achieve three weeks of continuous abstinence. 20% of patients on mirtazapine did not have any detectable blood level, therefore, poor compliance may have prevented detection of a medication effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes